CLINICAL TRIAL: NCT06930573
Title: A Single-Arm, Multicenter, Exploratory Clinical Study on the Efficacy and Safety of AK112 in Perioperative Treatment of Resectable Hepatocellular Carcinoma With High Recurrence Risk
Brief Title: A Study of AK112, a PD-1/ VEGF Bispecific Antibody, for Resectable Hepatocellular Carcinoma With High Recurrence Risk
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Zujiang YU, MD, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L2024-K001-006
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-02

CONDITIONS: HCC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Resectable Hepatocellular Carcinoma With High Recurrence Risk (Experimental)
  Interventions: Drug: AK112

INTERVENTIONS:
Drug: AK112 — After enrollment, patients receive AK112 at 20 mg/kg, administered via intravenous infusion on day 1 of each cycle, every 3 weeks (Q3W). After four cycles, surgery is performed four weeks after the last dose. AK112 at 20 mg/kg is administered again four to eight weeks after surgery, via intravenous infusion on day 1 of each cycle, every 3 weeks (Q3W), until disease progression, death, intolerable toxicity, withdrawal of consent, initiation of new anti-tumor therapy, or other reasons specified in the protocol for discontinuation of treatment. The maximum postoperative treatment duration with AK112 is 12 months.

SUMMARY:
This study is a single-arm, open-label study. To assess the efficacy and safety of AK112 therapy in patients with resectable hepatocellular carcinoma at high risk of recurrence. The primary endpoint is the 12-month RFS rate of resectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent before any trial-related procedures. 2. Male or female aged between 18 and 75 years. 3. ECOG PS score 0-1. 4. Histologically/cytologically confirmed hepatocellular carcinoma (HCC) or meets clinical diagnosis criteria (per 2022 Chinese Primary Liver Cancer Diagnosis and Treatment Guidelines).

5. No preoperative HCC treatment (including chemotherapy, targeted therapy, immunotherapy, cell therapy, local radiotherapy, ablation, or intervention). No lymph node invasion/distant metastasis on preoperative imaging, and deemed suitable for radical surgery by the investigator.

6. At least one postoperative high-risk factor for HCC recurrence:

1. Single lesion more than 5 cm in longest diameter.
2. Microvascular or macrovascular invasion.
3. More than 3 tumor nodules.
4. Edmondson grade at least II on tumor pathology.
5. AFP more than 400 μg/L in CNLC Ib-IIa patients.
6. Tumor adjacent to blood vessels in CNLC Ib-IIa patients.
7. Incomplete tumor capsule in CNLC Ib-IIa patients. 7. Child-Pugh score A or B7. 8. Expected survival more than 3 months. 9. At least one measurable lesion per RECIST 1.1. 10. Total T3 or free T3 and free T4 within normal range (thyroid replacement therapy allowed). Asymptomatic subjects with abnormal T3, free T3, or free T4 are eligible.

   11. Adequate organ and bone marrow function, with laboratory values meeting the following criteria within 7 days before randomization (no blood products, growth factors, albumin, or corrective treatments within 14 days before obtaining these results):
   1. Hematology: ANC at least 1.5×10⁹/L; PLT at least 75×10⁹/L; HGB at least 9.0 g/dL.
   2. Liver function: TBIL at most 3×ULN; ALT, AST, ALP at most 5×ULN; serum albumin at least 28 g/L.
   3. Renal function: Serum creatinine at most 1.5×ULN or CCr at least 50 mL/min (Cockcroft-Gault formula); urine protein less than 2+ on urinalysis. For subjects with baseline urine protein at least 2+, 24-hour urine protein less than 1 g.
   4. Coagulation: INR and APTT at most 1.5×ULN. 12. For female subjects of childbearing potential, a negative urine or serum pregnancy test within 3 days before the first study drug administration (Cycle 1, Day 1). If urine test is inconclusive, a blood pregnancy test is required. Postmenopausal females (for at least 1 year), surgically sterilized, or hysterectomized are not of childbearing potential.

   13. All subjects with pregnancy risk must use effective contraception throughout treatment until 120 days after the last study drug dose (or 180 days after last chemotherapy dose).

   Exclusion Criteria:
   1. Past histological/cytological diagnosis of fibrolamellar hepatocellular carcinoma (HCC), sarcomatoid HCC, cholangiocarcinoma, etc.
   2. Other malignancies within 5 years before enrollment, except those locally treated HCC. Exceptions include basal/squamous cell skin cancer, superficial bladder cancer, cervical/ breast carcinoma in situ.
   3. History of hepatic encephalopathy or liver transplantation.
   4. Cancer thrombus in portal vein branches, superior mesenteric vein, or inferior vena cava.
   5. Active hepatitis B/C infection, with HBV DNA more than 2000 IU/ml or 10⁴ copies/ml; HCV RNA more than 10³ copies/ml; co-positive HBsAg and anti-HCV. Those on antiviral therapy meeting the above criteria and willing to continue during the study are eligible.
   6. Clinically symptomatic pleural effusion, ascites, or pericardial effusion requiring drainage.
   7. Esophagogastric variceal bleeding due to portal hypertension within 6 months before first dose; current imaging shows significant esophagogastric varices.
   8. History of significant bleeding tendency/coagulopathy; clinically significant bleeding within 1 month before first dose (e.g., GI bleeding, hemoptysis, epistaxis); continuous antiplatelet/anticoagulant therapy within 10 days before first dose.
   9. Arterial/venous thromboembolism within past 6 months, including myocardial infarction, unstable angina, stroke, transient ischemic attack, pulmonary embolism, deep vein thrombosis. Exceptions: stable thrombosis after routine anticoagulation for implanted venous ports/ catheters or superficial vein thrombosis; low-dose LMWH (e.g., enoxaparin 40 mg/day) allowed.
   10. History of myocarditis, cardiomyopathy, malignant arrhythmias. Unstable angina, MI, CHF (NYHA ≥Class 2), or vascular disease requiring hospitalization within 12 months before first dose; other cardiac impairments affecting drug safety assessment. Severe ulcers, unhealed wounds, GI perforation, fistula, obstruction, abscess, or acute GI bleeding within 6 months before first dose; thromboembolic events, TIA, stroke within 6 months before first dose; COPD exacerbation, hypertensive crisis/encephalopathy within 1 month before first dose; current hypertension uncontrolled by oral medication (systolic BP more than 150 mmHg or diastolic BP more than 90 mmHg).
   11. History or current non-infectious pneumonia/interstitial lung disease requiring systemic corticosteroids; active or past definite inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, chronic diarrhea); active autoimmune disease requiring systemic treatment within past 2 years (e.g., DMARDs, corticosteroids, immunosuppressants). Replacement therapy (e.g., thyroid hormones, insulin, physiological corticosteroids for adrenal/pituitary insufficiency) is not considered systemic treatment.
   12. History of immunodeficiency; positive HIV antibody test; current long-term use of systemic corticosteroids or other immunosuppressants (except short-term corticosteroids for COPD-related dyspnea or temporary allergy prevention).
   13. Known active tuberculosis (TB); suspected active TB requires clinical exclusion; known active syphilis infection.
   14. Severe infection within 4 weeks before first dose (e.g., requiring hospitalization, sepsis, severe pneumonia); active infection treated with systemic anti-infectives within 2 weeks before first dose (excluding antiviral therapy for hepatitis B/C).
   15. Past systemic chemotherapy or bevacizumab/biosimilar treatment.
   16. Past immunotherapy, including immune checkpoint inhibitors (e.g., anti-PD-1/L1, CTLA-4, CD47, SIRPα, LAG-3 antibodies), immune checkpoint agonists (e.g., ICOS, CD40, CD137, GITR, OX40 antibodies), or any immunotherapy targeting tumor immune mechanisms.
   17. Past local therapy for liver lesions, including TACE, TARE, HAIC, or radiotherapy.
   18. Systemic anti-tumor traditional Chinese medicine or immunomodulatory drugs (e.g., thymosin, interferon, interleukin) within 2 weeks before first dose (except those locally used to control pleural/ascitic fluid).
   19. Live/attenuated vaccine administration within 30 days before first dose or planned during study; inactivated vaccines are allowed.
   20. Known allergy to any study drug component; history of severe hypersensitivity to other monoclonal antibodies.
   21. Known psychiatric disease, drug abuse, alcoholism, or substance addiction.
   22. Pregnant or breastfeeding women.
   23. Any condition, disease, or abnormality that may interfere with study results, hinder study participation, or pose additional risk, as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-05-24 (Estimated); Study Completion 2027-12-24 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 1 years
  Progression-free survival is defined as the time from the start of treatment with AK112 until the first documentation of disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No